CLINICAL TRIAL: NCT04454268
Title: Intracranial Hydatid Cyst: Series of 8 Cases
Brief Title: Intracranial Hydatid Cyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, ahmed salaheldin mohammed saro, Assistant professor of neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intracranial Hydatid Cyst
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hydatid cyst (Other)
  Interventions: Procedure: cyst extirpation

INTERVENTIONS:
Procedure: cyst extirpation — complete removal of the cyst without rupture

SUMMARY:
Central nervous system (CNS) hydatid cysts is a rare presentation of hydatid cyst, although may be the cause of intracranial space-occupying lesions in 4% in endemic countries. It affects mostly children. The diagnosis of CNS hydatid is still problematic in spite of the advancements in imaging techniques (CT or MRI). Extirpation of the intact cyst is the treatment of choice, resulting in most cases to a complete recovery.

DETAILED DESCRIPTION:
Hydatid disease is a parasitic induced disease caused by either Echinococcus granulosus or Echinococcus multilocularis during the larval stage of these tapeworms. Hydatid cysts are endemic in many countries, such as Latin America (Argentina, Brazil, Chile, Peru, and Uruguay); followed by Europe (France, Italy, and Greece), the Middle East (Turkey, Lebanon, Syria, and Jordan), Southeast Asia (China, Iran, and India) and Africa (Tunisia and less commonly, Egypt)

ELIGIBILITY:
Inclusion Criteria:

* intracranial hydatid cyst

Exclusion Criteria:

* Arachnoid cysts
* conservative treatment

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
number of patients who haven total removal of intracranial cyst | 7 years
  degree of consciousness incomplete extirpation without removal without neurological deficit 0 space